CLINICAL TRIAL: NCT04810533
Title: A Single-center, Open-label, Single-dose Phase I Study to Investigate the Absorption, Metabolism and Excretion of [14C]SH-1028 in Chinese Healthy Male Subjects
Brief Title: The Absorption, Metabolism and Excretion of [14C]SH-1028 in Chinese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SHC013-I-04
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — SH-1028

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C] SH-1028 (Experimental): Volunteers will receive 200 mg [14C] SH-1028 containing a nominal 88 μCi activity, administered by mouth, as a solution.
  Interventions: Drug: [14C] SH-1028

INTERVENTIONS:
Drug: [14C] SH-1028 — Volunteer will receive a single oral dose of 200 mg/88 uCi [14C]SH-1028 as a solution on Day 1

SUMMARY:
This is a single-center, open-label, single-dose phase I study to investigate the absorption, metabolism and excretion of [14C] SH-1028 in healthy Chinese male subjects. The study will be conducted into two steps：Firstly, 2 subjects are enrolled in to participate in the pilot study to grope for the collection time of plasma, urine and feces sampling post-dose. Then, the collection time of blood and excreta samples (urine and feces) from the subsequent 2-4 subjects will be adjusted according to the pilot study.

DETAILED DESCRIPTION:
Subjects who had signed informed consent and meet inclusion criteria and no exclusion criteria are admitted to Phase I Clinical Unit two days prior to dosing (D-2). On the morning of Day 1 before dosing, subjects will be transferred to nuclear medical ward. And after an overnight fast of at least 10 h, subjects will receive a single oral dose of 200 mg (88 μCi) of [14C]SH-1028 as an oral suspension. Then, after two days of the dosing, subjects will be transferred back to Phase I Clinical Unit ward and confined to this unit until blood or excreta sampling and safety monitoring at the designated time points or intervals are complete.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers between the age of 18 to 50 years old；
2. Body weight >=50 kg, Body mass index between 19 and 26 kg/m2 (including 19 and 26 kg/m2);
3. Normal physical findings, clinical laboratory values, vital signs and 12-lead ECG, or any abnormality that is non-clinically significant;
4. Male subjects of reproductive potential with partners will be instructed to, and must be willing to practice a highly effective method of birth control for the duration of the study and continuing 6 months after discontinuing treatment with the investigational product.;
5. Signing the informed consent forms by oneself;
6. Be able to communicate well with the researcher and be able to complete the trial in accordance with the program.

Exclusion Criteria:

1. History of or current clinically significant cardio, pulmonary, endocrine, metabolism, renal, hepatic, gastrointestinal, dermatology, infection, hematology, neurological, mental disease or disorder;
2. Positive test for HBs-Ag, HCV-Ab, HIV-Ab, or syphilis antibody;
3. Long-QT syndrome or family history of it, or QTcF interval > 450 mses;
4. Allergies, have allergies to drugs or foods; or have known allergies to the components of the drug;
5. Those who smoked daily >5 sticks of cigarette 3 months prior to first dose or cannot give up smoking during study；
6. The weekly alcohol consumption was higher than 14 units of alcohol (1 unit=10ml or 8g absolute alcohol. 25 ml 40% liquor, 330ml 5% beers, 175ml 12% grape wine are equal to 1.0, 1.5 and 2.0 units of alcohol respectively) 3 months prior to screening period, or positive test for the alcohol breath test results during screening period；
7. Those have history of drug abuse or taking soft drug (i.e., marihuana); or the results of urine test in drugs were positive;
8. Participated in other clinical trials within 3 months before screening;
9. Received any drug within 14 days before taking the investigational drug;
10. Received any drugs that inhibit or induce the CYP450 enzyme (i.e., inducers- barbiturates, tegretol, phenytoin, rifampicin, hexadecadrol, rifabutin, rifapentini; inhibitors- SSRI-antidepressant, cimetidine, diltiazem, macrolides, verapamil, imidazoles- antifungal drugs) 30 days prior to screening period；
11. History of syncope / needle syncope and intolerable intravenous indwelling needle;
12. Those who have undergone major surgery within the first 6 months of the screening period;
13. Those who have habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease；
14. Hemorrhoids or perianal disease with regular/perianal bleeding;
15. Significant radiation exposure within one year prior to drug administration (more than one exposure from chest X-ray, CT scan, or barium meal examination and radiation-related occupations);
16. Those who cannot complete this study because of other reasons, or any factors judged by investigator that the participants cannot meet.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
The percentage of radioactive dose of [14C] radiolabelled SH-1028 recovered in blood and in total, up to Day 15 | Blood samples : - 0.5hrs, 1hrs, 2hrs, 3hrs, 4hrs, 6hrs, 8hrs, 12hrs, 24hrs, 48hrs, 72hrs, 120hrs, 168hrs, 216hrs, 264hrs and 336hrs
  The distribution of [14C]SH-1028 in the whole blood and plasma and whole radioactive pharmacokinetics following the single orally administered [14C]SH-1028 in healthy male volunteers.
The percentage of radioactive dose of [14C] radiolabelled SH-1028 recovered in urine, faeces and in total, up to Day 15. | Day1 to Day 15
  Quantitive analysis of whole radioactivity of excrement of orally administered [14C]SH-1028 in healthy volunteers to obtain the mass balance data and the main excretion pathway in human body.
The concentrations of SH-1028, Imp2 and Imp3 in plasma up to Day 15 | Blood samples : - 0.5hrs, 1hrs, 2hrs, 3hrs, 4hrs, 6hrs, 8hrs, 12hrs, 24hrs, 48hrs, 72hrs, 120hrs, 168hrs, 216hrs, 264hrs and 336hrs
  Quantitive analysis of the concentrations of SH-1028 and Imp2,Imp3 (Metabolites of SH-1028) in plasma using the validated LC-MS/MS to obtain pharmacokinetic data.
Proportion of different metabolites | Blood samples : - 0.5hrs, 1hrs, 2hrs, 3hrs, 4hrs, 6hrs, 8hrs, 12hrs, 24hrs, 48hrs, 72hrs, 120hrs, 168hrs, 216hrs, 264hrs and 336hrs
  Proportion of different metabolites in healthy volunteers after oral administration of [14C]SH-1028
Types of adverse events | Baseline (Day-2) to Day 15
  Types of adverse events assessed by CTCAE v5.0 that occurred during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shao, Ph D, Principal Investigator — Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine; Wei Liu, M.A, Principal Investigator — Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine
Locations (1):
- Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No